CLINICAL TRIAL: NCT04339023
Title: Open-Label Placebo Treatment for Acute Postoperative Pain: A Randomized Controlled Trial (OLP-POP Study)
Brief Title: Open-Label Placebo Treatment for Acute Postoperative Pain
Acronym: OLP-POP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-00099;qu19Ruppen
Record Dates: First submitted 2020-03-21; First posted 2020-04-08 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Postoperative Pain
Keywords: postoperative pain; Open-Label Placebo; morphine; Transforaminal Lumbar Interbody Fusion
MeSH Terms: conditions — Pain, Postoperative | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OLP-Group (Experimental): patients will receive in addition to TAU, 2 open-label Placebo (OLP) injections (containing each 5 ml of NaCl 9%) per day for two consecutive days following minimally invasive TLIF
  Interventions: Drug: Open-Label Placebo
- TAU-group (Other): The treatment as usual (TAU) group will serve as control group and will control for the natural course of postoperative pain under usual medication intake, following minimally invasive TLIF
  Interventions: Other: treatment as usual

INTERVENTIONS:
Drug: Open-Label Placebo — in addition to Treatment as usual, patients receive placebos without concealment (open-label placebo, OLP)
  Arms: OLP-Group
Other: treatment as usual — usual medication intake following minimally invasive TLIF. TAU consists of 3 gram Paracetamol per os a day, a patient-controlled morphine pump (Maximum of 2 milligram (mg) every 12 minutes) and rescue medication (1000 mg of Metamizol, maximum every 6 hours)
  Arms: TAU-group

SUMMARY:
This study is to evaluate whether the amount of morphine intake in acute postoperative pain following minimally invasive Transforaminal Lumbar Interbody Fusion (TLIF) can be decreased with an Open-Label Placebo (OLP) intervention (comprising the administration of sodium chloride (NaCl) injections and an evidence-based treatment rationale) in comparison to a "Treatment As Usual" (TAU) control group.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Scheduled to receive a TLIF procedure at University Hospital Basel (USB)
* 18 years or older
* German speaking
* Able to understand the study and its outcome measures

Exclusion Criteria:

* Known chronic pain, which is unrelated to problem targeted by the surgery
* Known neuromuscular disease
* Known mental disorders
* Known drug or massive alcohol intake or of other psychoactive substances
* Known kidney or liver disease (glomerular filtration rate (GFR)/ GFR < 30)
* Contraindications to the class of drugs under investigation, e.g., known hypersensitivity or allergy to the investigational product
* Parallel participation in another study with investigational drugs
* More than 30 mg/day (equivalent dose of oral morphine) preoperative opioid consumption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Difference in morphine consumption | starting on the first day post-surgery at 09:00 am (T1) and ending on the third day of surgery at 09:00 am (T5). morphine records will be read out twice a day (9:00 am and 16:45)
  cumulative dose (i.e., total amount) of self-administered morphine within 48 hours starting on the first day post-surgery at 09:00 am (T1) and ending on the third day of surgery at 09:00 am (T5)

SECONDARY OUTCOMES:
Difference in morphine request rates | between T1 (9:00 am day post surgery) and T5 (9:00 am, 3rd day post surgery) (48 hours, morphine records will be read out twice a day (9:00 am and 16:45)
  Morphine demand behaviour will be measured by the total number of successful and unsuccessful clicks on the Patient Controlled Analgesia (PCA) pump between T1 and T5 (48 hours)
Difference in pain intensity at rest | The two "at rest" scales (for leg and back pain) will be administered every two hours starting after transport to normal ward on the day of surgery (T0) until 09:00 am on the third day post-surgery (T5) and as well before surgery (T-1)
  back and leg pain intensity at rest will be measured separately by two 11-point Numeric Rating Scales (NRS, i.e., back / leg pain intensity at rest), which assesses pain intensity by asking participants to rate their pain intensity on a 0 to 10 scale, where 0 is "no pain" and 10 is "worst pain possible"
Difference in pain intensity while walking | The two "while walking" scales will be administered the day before surgery (T-1), after transport to normal ward (i.e., at T0), at T2 (16:45, 1st day after surgery), T4 (16:45 2nd day post surgery), respectively.
  back and leg pain intensity while walking will be measured separately by two 11-point Numeric Rating Scales (i.e., back / leg pain intensity while walking), which assesses pain intensity by asking participants to rate their pain intensity on a 0 to 10 scale, where 0 is "no pain" and 10 is "worst pain possible"
Difference in comprehensive pain assessment and patients' perception of postoperative pain management | The scale will be administered on the day before surgery (T-1), in the morning of the first day post-surgery (i.e., between 07:00 and 09:00; T0) , after the pain nurse visit 09:00 am day 2 (T3) and 09:00 am day 3 (T5) post-surgery
  will be assessed by the German version of the International Pain Outcomes (IPO) Questionnaire. The IPO assesses patients pain experience and outcomes regarding patient reported aspects
Difference in requested rescue analgesics | After trial completion of participants, study team members will extract the data from hospital records for the time periods of: the day of surgery (T0) till first day post-surgery at 09:00 am (T1) and T1 to T5 (09:00 am day 3 post-surgery)
  will be regularly assessed as part of standard procedures of the hospital and will be documented in the electronic hospital record of each patient
Opioid-Related Side Effects | After trial completion of participants, study team members will extract the data from hospital records for the time periods of: the day of surgery (T0) till first day post-surgery at 09:00 am (T1) and T1 to T5 (09:00 am day 3 post-surgery)
  nausea, vomiting and constipation (i.e., stool frequency, vomiting and amount of delivered laxatives and antiemetics) are regularly assessed and documented as part of standard hospital procedures
Length of Post-Surgery Hospitalisation | Length of Post-Surgery Hospitalisation, approximately 14 days after surgery
  Length of Post-Surgery Hospitalisation, upon participants trial completion this data will be extracted by study team members from the electronic hospital record of each patient

CONTACTS AND LOCATIONS:
Overall Officials: Wilhelm Ruppen, Prof. Dr., Principal Investigator — University Hospital of Basel, Department of Anesthesia; Jens Gaab, Prof. Dr., Principal Investigator — University of Basel,Faculty of Psychology
Locations (1):
- University Hospital of Basel, Department of Anesthesia, Basel, Switzerland

REFERENCES:
- [Derived] Sezer D, de Leeuw M, Netzer C, Dieterle M, Meyer A, Buergler S, Locher C, Ruppen W, Gaab J, Schneider T. Open-Label Placebo Treatment for Acute Postoperative Pain (OLP-POP Study): Study Protocol of a Randomized Controlled Trial. Front Med (Lausanne). 2021 Nov 5;8:687398. doi: 10.3389/fmed.2021.687398. eCollection 2021. PMID 34805194